CLINICAL TRIAL: NCT02353312
Title: Rhode Island Diastolic Dysfunction - Heart Failure
Acronym: RIDD-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Collaborators: BioMarin Pharmaceutical (Industry); Lifespan (Other)
Responsible Party: Principal Investigator, Wen-Chih Wu, Staff Cardiologist, Providence VA Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-051
Record Dates: First submitted 2014-12-29; First posted 2015-02-02 (Estimated); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Cardiovascular Disease
Keywords: Diastolic; Biopterin; Therapeutic Use; Drug Therapy; Quality of Life
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Heart Murmurs | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial Intervention Arm (Experimental): Kuvan® supplementation in addition to standard care for heart failure for three months. At the end of three months, stop Kuvan®, patients will only receive Standard care for heart failure for another 3 months
  Interventions: Drug: Kuvan
- Delayed Intervention Arm (Active Comparator): Standard care for heart failure for three months. At the end of three months, Starting Kuvan® supplementation in addition to Standard care for heart failure for another 3 months
  Interventions: Drug: Kuvan

INTERVENTIONS:
Drug: Kuvan — Kuvan® (sapropterin dihydrochloride) will be initiated at 10mg/kg/day with meals for one week. After telephone contact on day 7, assuming no adverse effects are noted, the patient will be instructed to increase their daily dose to 20mg/kg/day with meals for the remainder of the 3 months.
  Other Names: sapropterin dihydrochloride

SUMMARY:
To study the hypothesis that treating patients with underlying diastolic dysfunction with oral Kuvan® (BH4, also known as tetrahydrobiopterin) in addition to current best practices will improve metabolic and echocardiographic diastolic function parameters.

DETAILED DESCRIPTION:
Congestive heart failure carries a significant epidemiologic and economic burden in today's healthcare system and is associated with increased morbidity and mortality in those affected.

There are approximately 5 million people in the United States with heart failure, and of those, nearly half have heart failure with preserved ejection fraction (HFpEF). HFpEF, also referred to as diastolic heart failure, is a clinical syndrome characterized by prolonged relaxation of the myocardium resulting in symptoms including dyspnea, edema, fatigue, and decreased exercise tolerance, which are clinically indistinguishable from the presentation of heart failure with reduced ejection fraction (HFrEF). The underlying mechanisms in diastolic dysfunction are not clearly elucidated, making targeted therapy a challenge. There are currently no FDA approved treatments for this syndrome, and multiple clinical trials have demonstrated that standard treatments for systolic heart failure are ineffective in treating diastolic dysfunction. One of the proposed underlying mechanisms of diastolic dysfunction is via the reduction of nitric oxide (NO), an endothelium-derived vasodilator that regulates blood pressure and regional blood flow. In 2010, Silberman et al. examined the effect of cardiac oxidation on nitric oxide and found that depletion of tetrahydrobiopterin (BH4), an essential cofactor in the production of nitric oxide, causes uncoupling of nitric oxide synthase, impaired relaxation of cardiac myocytes, and leads to subsequent diastolic dysfunction. The authors further went on to demonstrate that treatment with BH4 can improve diastolic dysfunction in a hypertensive mouse model as well as in isolated cardiac myocytes and may play a role in the treatment of HFpEF.

To the investigators' knowledge, the role of BH4 in treating diastolic dysfunction in human subjects has not been studied.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female U.S. Veteran patients over the age of eighteen, with echocardiographic findings of >= Grade 2 diastolic dysfunction [as per American Society of Echocardiography guidelines] and
2. Diagnosis of hypertension, diabetes, or heart failure in medical records.
3. Eligible subjects must be ambulatory (not dependent on any ambulatory assist devices including cane or walker).

Exclusion Criteria:

1. Any history of documented ejection fraction <50%
2. Significant COPD (defined as oxygen-dependent COPD)
3. Acute coronary syndrome within the past three months defined by EKG changes and biomarkers of myocardial necrosis (ie. elevated troponin) in the setting of chest pain or an anginal equivalent)
4. Presence of hypertrophic cardiomyopathy
5. Presence of infiltrative/restrictive cardiomyopathy
6. Echocardiographic evidence of moderate or severe aortic or mitral valve stenosis or regurgitation
7. Previously diagnosed phenylketonuria
8. End stage renal disease requiring hemodialysis
9. Pre-existing seizure disorder
10. Terminal illness (not including heart failure) with expected survival of one year or less
11. Females who are pregnant or breastfeeding. All females of child bearing age will undergo pregnancy testing prior to randomization.
12. Recent hospitalization within three months.
13. Previous Bioprosthetic and/or mechanical aortic or mitral valves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chih Wu, MD, MPH, Principal Investigator — Providence VA Medical Center
Locations (1):
- Providence VAMC, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Kuvan First, Then no Kuvan: Kuvan® supplementation in addition to standard care for heart failure for three months. At the end of three months, stop Kuvan®, patients will only receive Standard care for heart failure for another 3 months
  Kuvan: Kuvan® (sapropterin dihydrochloride) will be initiated at 10mg/kg/day with meals for one week. After telephone contact on day 7, assuming no adverse effects are noted, the patient will be instructed to increase their daily dose to 20mg/kg/day with meals for the remainder of the 3 months.
- No Kuvan First, Then Kuvan: Standard care for heart failure for three months. At the end of three months, Starting Kuvan® supplementation in addition to Standard care for heart failure for another 3 months
  Kuvan: Kuvan® (sapropterin dihydrochloride) will be initiated at 10mg/kg/day with meals for one week. After telephone contact on day 7, assuming no adverse effects are noted, the patient will be instructed to increase their daily dose to 20mg/kg/day with meals for the remainder of the 3 months.
Period: Overall Study
Arm/Group | Kuvan First, Then no Kuvan | No Kuvan First, Then Kuvan
Started | 16 | 12
Completed | 13 | 10
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kuvan First, Then no Kuvan | No Kuvan First, Then Kuvan | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (9.78) | 72.1 (5.85) | 71.4 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Oxygen Consumption During Maximal Bike Exercise
Description: The change from baseline in oxygen consumption during maximal bike exercise. This was measured using cardiopulmonary exercise tress test (CPET), recorded in milliliters per kilogram per minute (mL/kg/min). Higher oxygen consumption scores indicate better aerobic capacity and cardiovascular function. An increase in oxygen consumption from baseline to post-intervention signifies an improvement in these areas. Conversely, a decrease would indicate a decline in aerobic capacity and cardiovascular health.
Time Frame: Baseline (period 0), 3 mos (period 1), 6 mos (period 2)
Population: All patients who had both baseline and final test.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Groups:
- On Kuvan: Kuvan® supplementation in addition to standard care for heart failure in either the first or last three months. Kuvan® (sapropterin dihydrochloride) will be initiated at 10mg/kg/day with meals for one week. After telephone contact on day 7, assuming no adverse effects are noted, the patient will be instructed to increase their daily dose to 20mg/kg/day with meals for the remainder of the 3 months.
- Not on Kuvan: Standard care for heart failure in either the first or last three months.
Arm/Group | On Kuvan | Not on Kuvan
Number analyzed (Participants) | 20 | 22
mL/kg/min | 14.45 (5.00) | 14.18 (3.69)
Statistical Analysis 1: Comparison: On Kuvan vs Not on Kuvan; Test type: Equivalence — Pairwise comparisons of VO2 max means with equal variances between participant on and off treatment; p = 0.823, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Description: There were 28 patients enrolled.
Groups:
- On Kuvan: Kuvan® supplementation in addition to standard care for heart failure for three months. At the end of three months, stop Kuvan®, patients will only receive Standard care for heart failure for another 3 months
  Kuvan: Kuvan® (sapropterin dihydrochloride) will be initiated at 10mg/kg/day with meals for one week. After telephone contact on day 7, assuming no adverse effects are noted, the patient will be instructed to increase their daily dose to 20mg/kg/day with meals for the remainder of the 3 months.
- Off Kuvan: Standard care for heart failure for three months. At the end of three months, Starting Kuvan® supplementation in addition to Standard care for heart failure for another 3 months
Arm/Group | On Kuvan | Off Kuvan
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 4/28 | 6/28
Other Adverse Events (participants affected / at risk) | 28/28 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On Kuvan (N=28) | Off Kuvan (N=28)
Hospitalizations (Investigations) | 2 (2) | 3 (3)
ER visit (Investigations) | 2 (2) | 3 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On Kuvan (N=28) | Off Kuvan (N=28)
Fever (Infections and infestations) | 1 (2) | 3 (5)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (3)
Emesis (Gastrointestinal disorders) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 12 (20) | 8 (17)
Rhinorrhea (Blood and lymphatic system disorders) | 14 (17) | 7 (8)
weight gain (General disorders) | 12 (19) | 12 (16)
JVD (Vascular disorders) | 4 (5) | 6 (6) — Jugular venous distension
Pulmonary crackles (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Peripheral abdominal edema (Vascular disorders) | 21 (34) | 16 (27)
Other (Vascular disorders) | 15 (21) | 17 (25)

LIMITATIONS AND CAVEATS:
Incomplete or missing data for only seven participants leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT02353312/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT02353312/ICF_001.pdf